CLINICAL TRIAL: NCT01156662
Title: Efficacy of Thrombosuction in Primary Percutaneous Coronary Intervention of Acute Myocardial Infarction
Acronym: ETAMI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ajou University School of Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Seung-Jea Tahk, Dr., Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETAMI-2009
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Thrombus aspiration; Percutaneous coronary intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No aspiration (Active Comparator)
  Interventions: Device: Endeavor resolute or Resolute integrity (Medtronic)
- Thrombus aspiration (Active Comparator)
  Interventions: Device: Export Aspiration Catheter, Endeavor resolute or Resolute integrity (Medtronic)

INTERVENTIONS:
Device: Endeavor resolute or Resolute integrity (Medtronic) — PCI without thrombus aspiration
  Arms: No aspiration
Device: Export Aspiration Catheter, Endeavor resolute or Resolute integrity (Medtronic) — PCI after thrombus aspiration
  Arms: Thrombus aspiration

SUMMARY:
The present study was designed to investigate whether the thrombus aspiration using Export Aspiration Catheter (Medtronic Corporation, California, USA) during primary percutaneous coronary intervention (PCI) in acute myocardial infarction improve clinical outcomes.

DETAILED DESCRIPTION:
Primary percutaneous coronary intervention (PCI) is the preferred strategy for immediate revascularization in patients with acute ST-elevation myocardial infarction (STEMI). A meta-analysis of trials comparing primary PCI to fibrinolytic therapy showed a mortality benefit to the invasive approach. However, although TIMI III flow is achieved in the culprit epicardial vessel in the majority of patients, lack of tissue-level reperfusion is observed in approximately 30% of patients as manifested by persistence of chest pain and ST-segment elevation. Many strategies have tried to overcome this problem, from mechanical thrombectomy and distal protection devices to myocardial preserving agents. The purpose of present study is to investigate the efficacy of the thrombus aspiration using Export Aspiration Catheter (Medtronic Corporation, California, USA) during primary PCI in acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first ST-elevation myocardial infarction who undergo primary PCI within 12 hours after symptom onset
* Patients who are eligible for PCI

Exclusion criteria

* History of bleeding diathesis or coagulopathy
* Pregnant
* Known hypersensitivity or contra-indication to contrast agent
* Left main disease
* In-stent restenosis lesion
* Graft vessels lesion
* Chronic total occlusion lesion
* Renal dysfunction, creatinine more than 2.0 mg/dL
* Contraindication to aspirin, clopidogrel or cilostazol
* Prior PCI or bypass surgery
* Old myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2009-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The composite of cardiac death, Q-wave myocardial infarction, and target vessel revascularization | 12 months after index procedure

SECONDARY OUTCOMES:
All-cause Death | 1 month until 12 months after index procedure
Cardiac death | 1 month until 12 months after index procedure
Myocardial infarction(Q or non-Q) | 1 month until 12 months after index procedure
Stent thrombosis by Academic Research Consortium definition | 1 month until 12 months after index procedure
Target vessel revascularization (clinically- and ischemia-driven) | 1 month until 12 months after index procedure
Target lesion revascularization (clinically- and ischemia-driven) | 1 month until 12 months after index procedure
Post-procedural Thrombolysis in Myocardial Infarction (TIMI) flow grade | Day 0 (during PCI procedure)
Post-procedural Thrombolysis in Myocardial Infarction Myocardial Perfusion (TMP) grades | Day 0 (during PCI procedure)
Left ventricular wall motion improvement | 12 months
ST segment resolution on ECG after procedure | 0 hour (at the end of procedure), 1 hour, and 24 hours after PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jea Tahk, MD, PhD, Principal Investigator — Department of Cardiology, Ajou University School of Medicine, Ajou University Medical Center
Locations (27):
- South Korea (27):
  - Hallym University Sacred Heart Hospital, Anyang
  - Sejong General Hospital, Bucheon-si
  - Bundang CHA General Hospital, Bundang
  - Seoul National University Bundang Hospital, Bundang
  - Dankook University Hospital, Cheonan
  - Soon Chun Hyang University Hospital, Cheonan
  - Keimyung University Dongsan Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daejeon ST. Mary's Hospital,The Catholic University of Korea, Daejeon
  - Konyang University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Kwandong University college of Medicine Myongji Hospital, Goyang
  - National Health Insurance Corporation ILSAN Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Handong University Sunlin Hospital, Pohang
  - Inje University Pusan Paik Hospital, Pusan
  - Hallym University Kangdong Sacred Heart Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea Univeristy Guro Hospital, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - St. Carollo Hospital, Suncheon
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan
  - Yeonsei Univeristy Wonju College of Medicine Wonju Christion Hospital, Wŏnju